CLINICAL TRIAL: NCT01513902
Title: An Open-label Multiple Dose Study To Evaluate The Pharmacokinetics, Safety And Tolerability Of CP-690,550 In Pediatric Patients From 2 To Less Than 18 Years Of Age With Juvenile Idiopathic Arthritis (JIA)
Brief Title: Pharmacokinetics Of CP-690,550 In Pediatric Patients With Juvenile Idiopathic Arthritis (JIA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A3921103; 2011-004914-40 (EudraCT Number)
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Results first posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-05

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Arthritis; Pediatric; Tofacitinib; JIA
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Ages 12 to less than 18
  Interventions: Drug: CP-690,550
- Cohort 2 (Experimental): Ages 6 to less than 12
  Interventions: Drug: CP-690,550
- Corhort 3 (Experimental): Ages 2 to less than 6
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — CP-690,550 will be administered orally twice daily according to the dosing regimen provided below. Oral solution will be used for children weighing <40 kg. Oral tablets will be used for children weighing ≥40 kg. Children aged 12 to less than 18 years who are unable to swallow tablets will have the option of taking oral solution. Body Weight (kg) Dose (mg) Volume (mL) 5-11 1 1; 12-18 1.5 1.5; 19-24 2 2; 25-31 2.5 2.5; 32-39 3 3; ≥40 5 5
  Other Names: Tofacitinib
  Arms: Cohort 1
Drug: CP-690,550 — CP-690,550 will be administered orally twice daily according to the dosing regimen provided below. Oral solution will be used for children weighing <40 kg. Oral tablets will be used for children weighing ≥40 kg. Children less than 12 years of age with a body weight of ≥40 kg will have the option of taking oral solution or tablets. Body Weight (kg) Dose (mg) Volume (mL) 5-11 1 1; 12-18 1.5 1.5; 19-24 2 2; 25-31 2.5 2.5; 32-39 3 3; ≥40 5 5
  Other Names: Tofacitinib
  Arms: Cohort 2
Drug: CP-690,550 — CP-690,550 will be administered orally twice daily according to the dosing regimen provided below. Children with a body weight ≥30 kg will have the option of taking oral solution or tablets, and children weighing <30 kg will be dosed with the oral solution. Body Weight (kg) Dose (mg) Volume (mL) 5-6 1 1; 7-9 1.5 1.5; 10-12 2 2; 21-15 2.5 2.5; 16-19 3 3; 20-22 3.5 3.5; 23-26 4 4; 27-29 4.5 4.5; ≥30 5 5
  Other Names: Tofacitinib
  Arms: Corhort 3

SUMMARY:
Phase 1 study to describe pharmacokinetics of CP-690,550 in pediatric patients 2 to less than 18 years of age with Juvenile Idiopathic Rheumatoid Arthritis (JIA).

DETAILED DESCRIPTION:
This is an open-label, non-randomized, multi-center, oral CP-690,550, multiple-dose (twice daily for 5 days [except Day 5 when only morning dose will be given]) study in pediatric subjects with JIA aged from 2 to less than 18 years. Baseline visit will occur within 1 month of the completion of the Screening Visit. The study will consist of three cohorts based on the age of the subjects, Cohort 3: 2 to less than 6 years, Cohort 2: 6 to less than 12 years and Cohort 1: 12 to less than 18 years. In each cohort, at least 8 pediatric subjects with JIA will participate in the study ensuring a total number of at least 24 pediatric evaluable subjects completing the PK period.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients with JIA aged from 2 to less than 18 years with active JIA (extended oligoarthritis, polyarthritis rheumatoid factor positive or negative, psoriatic arthritis, enthesitis related arthritis), in 5 or more joints (using American College Rheumatology definition of active joint) at the time of the first study drug administration.
2. For subjects receiving MTX treatment, minimum duration of therapy is 4 months and dose stable for at least 6 weeks prior to first dose of study drug. MTX may be administered either orally or parenterally at doses not to exceed 20 mg/wk or 15 mg/m2/week.
3. A negative QuantiFERON-TB Gold In-Tube test performed within the 3 months prior to screening. A negative PPD test can be substituted for the QuantiFERON-TB Gold In-Tube test only if the central laboratory is unable to perform the test or cannot determine the results to be positive or negative and the Pfizer medical monitor approves it, on a case-by-case basis.

Exclusion Criteria:

1. Systemic JIA, persistent oligoarthritis, undifferentiated arthritis.
2. Current or recent history of uncontrolled clinically significant renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, or neurological disease.
3. History of any other rheumatic autoimmune disease.
4. Infections:

   1. Latent or active TB or any history of previous TB.
   2. Chronic infections.
   3. Any infection requiring hospitalization, parenteral antimicrobial therapy or judged to be opportunistic by the investigator within the 6 months prior to the first dose of study drug.
   4. Any treated infections within 2 weeks of Baseline visit.
   5. A subject known to be infected with human immunodeficiency virus (HIV), hepatitis B or hepatitis C virus.
   6. History of infected joint prosthesis with prosthesis still in situ.
5. History of recurrent (more than one episode) herpes zoster or disseminated (a single episode) herpes zoster or disseminated (a single episode) herpes simplex.
6. The biologic agents and DMARDs are disallowed at any time during this study. If a subject needs to be treated with one of these agents, the subject should be discontinued from the study.
7. Subjects who have been vaccinated with live or attenuated vaccines within the 6 weeks prior to the first dose of study medication or is to be vaccinated with these vaccines at any time during treatment or within 6 weeks following discontinuation of study drug.
8. Subjects with a malignancy or with a history of malignancy with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (4):
  - Explorer Clinic, University of Minnesota Children's Hospital, Minneapolis, Minnesota
  - Clinical and Translational Science Institute Masonic Clinical Research Unit (Administration Only), Minneapolis, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Randall Children's Hospital at Legacy Emanuel, Portland, Oregon
- Germany (3):
  - PRI - Pediatric Rheumatology Research Institute GmbH, Bad Bramstedt
  - Hamburger Zentrum fuer Kinder-und Jugendrheumatologie SchoenKlinik Hamburg Eilbek, Hamburg
  - Asklepios Klinik Sankt Augustin Gmbh, Sankt Augustin
- Poland (2):
  - Wojewodzki Specjalistyczny Szpital Dzieciecy im. Sw. Ludwika w Krakowie, Krakow
  - Klinika Kardiologii i Reumatologii Dzieciecej, Lodz
- Narodny ustav reumatickych chorob, Piešťany, Slovakia

REFERENCES:
- [Derived] Chang C, Vong C, Wang X, Hazra A, Diehl A, Nicholas T, Mukherjee A. Tofacitinib pharmacokinetics in children and adolescents with juvenile idiopathic arthritis. CPT Pharmacometrics Syst Pharmacol. 2024 Apr;13(4):599-611. doi: 10.1002/psp4.13104. Epub 2024 Jan 31. PMID 38298058
- [Derived] Ruperto N, Brunner HI, Zuber Z, Tzaribachev N, Kingsbury DJ, Foeldvari I, Horneff G, Smolewska E, Vehe RK, Hazra A, Wang R, Mebus CA, Alvey C, Lamba M, Krishnaswami S, Stock TC, Wang M, Suehiro R, Martini A, Lovell DJ; Pediatric Rheumatology International Trials Organization (PRINTO); Pediatric Rheumatology Collaborative Study Group (PRCSG). Pharmacokinetic and safety profile of tofacitinib in children with polyarticular course juvenile idiopathic arthritis: results of a phase 1, open-label, multicenter study. Pediatr Rheumatol Online J. 2017 Dec 28;15(1):86. doi: 10.1186/s12969-017-0212-y. PMID 29282090
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921103&StudyName=Pharmacokinetics%20Of%20CP-690%2C550%20In%20Pediatric%20Patients%20With%20Juvenile%20Idiopathic%20Arthritis%20%28JIA%29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants aged 2 to less than (<)18 years with juvenile idiopathic arthritis (JIA) were enrolled in the study.
Groups:
- Cohort I: 12 Years to <18 Years: CP-690,550 was administered orally, twice daily as oral solution (ranging from 1 milliliter [mL] to 3 mL) for children weighing <40 kilogram (kg) or twice daily as oral tablets (5 milligram [mg]) for participants weighing greater than or equal to (>=) 40 kg. Participants who were unable to swallow tablets had the option of taking oral solution.
- Cohort II: 6 Years to <12 Years: CP-690,550 was administered orally, twice daily as oral solution (ranging from 1 mL to 3 mL) for participants weighing <40 kg, oral tablets (5 mg) were used for participants weighing >=40 kg. Participants with a body weight of >=40 kg had the option of taking oral solution (5 mL) or tablets (5 mg).
- Cohort III: 2 Years to <6 Years: CP-690,550 was administered orally, twice daily as oral solution (ranging from 1 mL to 4.5 mL) for participants weighing <30 kg. Participants weighing >=30 kg had the option of taking oral solution (5 mL) or tablets (5 mg).
Period: Overall Study
Arm/Group | Cohort I: 12 Years to <18 Years | Cohort II: 6 Years to <12 Years | Cohort III: 2 Years to <6 Years
Started | 8 | 9 | 9
Completed | 8 | 9 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis population included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I: 12 Years to <18 Years | Cohort II: 6 Years to <12 Years | Cohort III: 2 Years to <6 Years | Total
Number analyzed (Participants) | 8 | 9 | 9 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (2.0) | 9.4 (1.8) | 4.0 (1.0) | 9.0 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 7 | 17
  Male | 3 | 4 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Apparent Oral Clearance (CL/F)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is also influenced by the fraction of the dose absorbed. Clearance was estimated by non compartmental analysis (NCA) of PK data. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. It was calculated by dividing the given oral dose by AUCtau. AUCtau is the area under the plasma concentration time-curve from time zero to end of dosing interval.
Time Frame: Day 5: Pre-dose, 0.5, 1, 2, 4, 8 hours post dose
Population: The PK analysis population included all enrolled and treated participants who had at least 1 of the PK parameters of primary interest. Here 'number of participants analyzed (N)' signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Cohort I: 12 Years to <18 Years | Cohort II: 6 Years to <12 Years | Cohort III: 2 Years to <6 Years
Number analyzed (Participants) | 8 | 8 | 9
liter per hour | 28.09 (22) | 25.48 (40) | 20.53 (33)

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) All Causalities
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment emergent AEs included both serious and non-serious AEs.
Time Frame: Baseline up to 28 days after the last dose of study drug (Day 5)
Population: The safety analysis population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort I: 12 Years to <18 Years | Cohort II: 6 Years to <12 Years | Cohort III: 2 Years to <6 Years
Number analyzed (Participants) | 8 | 9 | 9
participants
  AE | 1 | 1 | 2
  SAE | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Participants with laboratory test abnormalities of potential clinical concern without regard to baseline abnormality were reported. Criteria: Hematology(hemoglobin,hematocrit,red blood cell[RBC] count:<0.8*lower limit of normal [LLN], platelets:<0.5*LLN/greater than [>]1.75*upper limit of normal[ULN], white blood cell [WBC] count:<0.6*LLN></0>1.5*ULN, lymphocytes, total neutrophils:<0.8*LLN or >1.2*ULN, basophils, eosinophil, monocytes:>1.2*ULN); Liver Function (total bilirubin: >1.5*ULN, aspartate aminotransferase,alanine aminotransferase, alkaline phosphatase:>3.0*ULN, total protein, albumin:<0.8*LLN or >1.2*ULN);Renal Function (blood urea nitrogen, creatinine:>1.3*ULN, uric acid:>1.2*ULN); Electrolytes (sodium:<0.95*LLN or >1.05*ULN,potassium,chloride,calcium,bicarbonate:<0.9*LLN or >1.1*ULN);Clinical chemistry (glucose <0.6*LLN or >1.5*ULN, creatine kinase:>3.0*ULN); Urinalysis (Urine WBC and RBC: greater than or equal to [>=] 6/High Power Field [HPF]).
Time Frame: Baseline up to Day 5
Population: The safety analysis population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort I: 12 Years to <18 Years | Cohort II: 6 Years to <12 Years | Cohort III: 2 Years to <6 Years
Number analyzed (Participants) | 8 | 9 | 9
participants | 3 | 1 | 5

4. Primary Outcome: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Criteria for vital signs of potentially clinical concern included supine/sitting pulse rate of <40 beats per minute (bpm) or >120 bpm, standing pulse rate of <40 bpm or >140 bpm, systolic blood pressure of >=30 millimeters of mercury (mmHg) change from baseline and systolic blood pressure <90 mmHg, diastolic blood pressure >=20 mmHg change from baseline and diastolic blood pressure <50 mm Hg.
Time Frame: Baseline up to Day 5
Population: The safety analysis population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort I: 12 Years to <18 Years | Cohort II: 6 Years to <12 Years | Cohort III: 2 Years to <6 Years
Number analyzed (Participants) | 8 | 9 | 9
participants | 0 | 0 | 0

5. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau)
Time Frame: Day 5: Pre-dose, 0.5, 1, 2, 4, 8 hours post dose
Population: The PK analysis population included all enrolled and treated participants who had at least 1 of the PK parameters of primary interest. Here 'N' signifies those participants who were analyzed for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Cohort I: 12 Years to <18 Years | Cohort II: 6 Years to <12 Years | Cohort III: 2 Years to <6 Years
Number analyzed (Participants) | 8 | 8 | 9
nanogram*hour per milliliter (ng*hr/mL) | 156.6 (25) | 118.8 (27) | 142.5 (32)

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Day 5: Pre-dose, 0.5, 1, 2, 4, 8 hours post dose
Population: The PK analysis population included all enrolled and treated participants who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort I: 12 Years to <18 Years | Cohort II: 6 Years to <12 Years | Cohort III: 2 Years to <6 Years
Number analyzed (Participants) | 8 | 9 | 9
nanogram per milliliter (ng/mL) | 46.97 (40) | 41.67 (29) | 66.15 (28)

7. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: Day 5: Pre-dose, 0.5, 1, 2, 4, 8 hours post dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort I: 12 Years to <18 Years | Cohort II: 6 Years to <12 Years | Cohort III: 2 Years to <6 Years
Number analyzed (Participants) | 8 | 9 | 9
hours | 0.750 (25) [0.500 to 6.90] | 1.00 (27) [0.500 to 2.05] | 0.500 (32) [0.500 to 1.92]

8. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Day 5: Pre-dose, 0.5, 1, 2, 4, 8 hours post dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Cohort I: 12 Years to <18 Years | Cohort II: 6 Years to <12 Years | Cohort III: 2 Years to <6 Years
Number analyzed (Participants) | 7 | 8 | 9
liter | 104.9 (35) [0.500 to 6.90] | 71.0 (40) [0.500 to 2.05] | 51.44 (34) [0.500 to 1.92]

9. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Day 5: Pre-dose, 0.5, 1, 2, 4, 8 hours post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort I: 12 Years to <18 Years | Cohort II: 6 Years to <12 Years | Cohort III: 2 Years to <6 Years
Number analyzed (Participants) | 7 | 8 | 9
hours | 2.616 (0.454) | 1.949 (0.294) | 1.771 (0.406)

10. Secondary Outcome: Taste Assessment
Description: Participants were evaluated for taste assessment using a 5 categories questionnaire. Participants were asked to answer one of the following to describe the taste of oral solution of tofacitinib: Dislike very much, dislike a little, not sure, like a little, or like very much. The taste assessment was only performed for participants who received the oral solution. Number of participants within each category are reported.
Time Frame: Day 1, Day 5
Population: The analysis population was defined as all participants who had received at least 1 oral solution formulation of tofacitinib.
Measure: Number; unit: participants
Arm/Group | Cohort I: 12 Years to <18 Years | Cohort II: 6 Years to <12 Years | Cohort III: 2 Years to <6 Years
Number analyzed (Participants) | 2 | 7 | 9
participants
  Day 1: Dislike very much | 0 (0.45350) | 1 (0.29396) | 1 (0.40634)
  Day 1: Dislike a little | 0 | 0 | 2
  Day 1: Not sure | 1 | 1 | 1
  Day 1: Like a little | 1 | 3 | 1
  Day 1: Like very much | 0 | 2 | 4
  Day 5: Dislike very much | 0 | 1 | 0
  Day 5: Dislike a little | 1 | 0 | 3
  Day 5: Not sure | 1 | 2 | 1
  Day 5: Like a little | 0 | 2 | 2
  Day 5: Like very much | 0 | 2 | 3

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after the last dose of study drug (Day 5)
Arm/Group | Cohort I: 12 Years to <18 Years | Cohort II: 6 Years to <12 Years | Cohort III: 2 Years to <6 Years
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/8 | 1/9 | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I: 12 Years to <18 Years (N=8) | Cohort II: 6 Years to <12 Years (N=9) | Cohort III: 2 Years to <6 Years (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.